CLINICAL TRIAL: NCT06603662
Title: Systemic Oral Glucocorticoids for the Treatment of Acute Osteoarthritis Pain in the Emergency Department
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2207448
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis; Osteoarthritis (OA) of the Knee; Osteoarthritis (OA) of the Shoulder; Osteoarthritis (OA) of the Hip
Keywords: osteoarthritis; acute pain; glucocorticosteroids; emergency department
MeSH Terms: conditions — Osteoarthritis; Acute Pain; Emergencies | interventions — Prednisone; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention A - Prednisone (Active Comparator): Subjects assigned to the Intervention A group will receive prednisone 50 mg once a day for 5 days, plus ibuprofen 600 mg every 8 hours for 5 days.
  Interventions: Drug: Prednisone
- Intervention B - Dexamethasone (Active Comparator): Subjects assigned to the Intervention B group will receive a single dose of dexamethasone 10 mg, plus ibuprofen 600 mg every 8 hours for 5 days.
  Interventions: Drug: Dexamethasone
- Control - Placebo (Placebo Comparator): Subjects assigned to the Control group will receive placebo once a day for 5 days, plus ibuprofen 600 mg every 8 hours for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Subjects assigned to the Intervention A group will receive oral prednisone 50 mg once a day for 5 days, plus standard ibuprofen 600 mg every 8 hours for 5 days.
  Arms: Intervention A - Prednisone
Drug: Dexamethasone — Subjects assigned to the Intervention B group will receive a single oral dose of dexamethasone 10 mg, plus standard ibuprofen 600 mg every 8 hours for 5 days.
  Arms: Intervention B - Dexamethasone
Drug: Placebo — Subjects assigned to the Control group will receive oral placebo once a day for 5 days, plus standard ibuprofen 600 mg every 8 hours.
  Arms: Control - Placebo

SUMMARY:
The purpose of this clinical trial is to compare the analgesic effects (relief of pain) of glucocorticoids (steroids) and pain medication versus pain medication alone in adult patients presenting to the emergency department with joint pain due to osteoarthritis. Steroids are drugs that can reduce inflammation and are used commonly for many different medical conditions.

In brief, the central aims of the study are to:

1. Assess the efficacy of adding oral glucocorticoid medications to the standard pain medications used to treat the pain of osteoarthritis.
2. Assess the safety and tolerability of oral glucocorticoid medication for the short-term treatment of osteoarthritis pain.

We hypothesize that: 1) The addition of glucocorticoids to standard pain medications will improve reported pain scores at 3 days following the initiation of treatment compared to standard pain medications alone and 2) The use of glucocorticoids will be well tolerated.

Participants in the study will be randomized (like flipping a coin) into one of three groups:

1. Study Group 1 (Control) receiving placebo pills (no active ingredient) once a day for 5 days, plus ibuprofen (pain medication) for 5 days.
2. Study Group 2 (Intervention A) who will receive prednisone (steroid) once a day for 5 days, plus ibuprofen (pain medication) for 5 days.
3. Study Group 3 (Intervention B) who will receive one dose of dexamethasone (steroid) followed by placebo pills (no active ingredient) once a day for 4 days, plus ibuprofen (pain medication) for 5 days.

In all groups, acetaminophen (a different pain medication) can be taken as needed for pain that is not controlled with ibuprofen.

Participants will:

* Receive follow up phone calls at 1, 3, 7 and 14 days.
* Report pain scores related to joint pain.
* Report the number of pills taken of the various medications used in the study.
* Report any adverse events incurred during the follow up period.

DETAILED DESCRIPTION:
BACKGROUND

Osteoarthritis (OA) constitutes a significant disease burden both within the United States (US) and globally. Recent data shows that upwards of 527 million people worldwide were affected by OA in 2019. Data from 2001-2005 suggests that over 77 million ambulatory visits in the US were attributed to arthritic and rheumatological disorders, of which OA was the predominant etiology. Patients often present to the emergency department (ED) with complaints of acute pain related to OA.

Current guidelines recommend both lifestyle interventions and pharmacological interventions for the treatment of OA-related pain. Oral non-steroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen, ketorolac, and diclofenac remain first-line agents for the treatment of OA-related pain with strong recommendations for this intervention from the American College of Rheumatology/ Arthritis Foundation. In contrast, the evidence for topical NSAID use for the treatment of OA pain is inconsistent regarding their benefit.

Glucocorticosteroids, or glucocorticoids, are commonly used for their anti-inflammatory effects. Intraarticular glucocorticoid injections are a recommended adjunct treatment for OA-related pain refractory to NSAIDs. The majority of clinical practice guidelines support their use in OA with recent data showing significant improvement in pain scores following intraarticular glucocorticoid injections. Although commonly used in the outpatient setting, intraarticular injections for OA are used less frequently in the ED. This is due to the time required to perform the procedure, the need for subsequent follow-up, and technical considerations.

Compared to oral administration, intraarticular glucocorticoid injections have less systemic absorption and the potential for decreased adverse effects; however, oral glucocorticoid regimens have been shown to be well tolerated when given in short courses for acute pain. A Cochrane review examining short-term oral glucocorticoid use for the treatment of radicular low back pain found no association with significant adverse effects, including hyperglycemia.

The use of glucocorticoid injections in OA has been studied robustly, but there has been very little research examining the utility of oral systemic glucocorticoids in the treatment of acute OA-related pain. The current literature is largely limited to OA specifically affecting the hand and does not include ED patients. Dossing et al. found that oral corticosteroids were effective in improving pain, functional status, and quality of life in patients with hand OA when compared to placebo. Similarly, a systematic review noted that oral glucocorticoid use for the treatment of hand OA reduced pain and improved functional status at 4-6 weeks. Dorleijn et al. did not study oral glucocorticoids specifically, but noted that intramuscular injections of glucocorticoids were more effective when compared to placebo for the reduction of negative symptoms in hip OA at 2 weeks and beyond. Surprisingly, no such positive results were observed with intraarticular glucocorticoid injections.

We aim to examine the effectiveness and safety of adding short-term oral systemic glucocorticoids to a standardized NSAID regimen in adult ED patients presenting with acute pain due to OA.

OBJECTIVES

1. Assess the efficacy of adding oral glucocorticoids (prednisone or dexamethasone) to the standard treatment of acute OA pain with NSAIDs.
2. Assess the safety and tolerability of systemic oral glucocorticoids for the short-term treatment of acute OA pain in ED patients.

We hypothesize the combination of oral glucocorticoids and NSAIDs will result in improved pain control for acute OA pain compared to NSAIDs alone and will be well tolerated.

STUDY DESIGN

This will be a randomized, controlled, single-blinded, superiority trial consisting of adult patients presenting to the WellSpan York Hospital ED with acute, large joint monoarticular pain related to underlying OA. Informed consent will be obtained by a member of the study team prior to data collection or study procedures.

Patients enrolled in the study will be randomized into one of three groups in a 1:1:1 ratio. Group 1 (control) will receive ibuprofen 600 mg every 8 hours, plus a placebo (no active ingredient) pill daily x 5 days. Group 2 (intervention A) will receive ibuprofen 600 mg every 8 hours, plus prednisone 50 mg daily x 5 days. Group 3 (intervention B) will receive ibuprofen 600 mg every 8 hours x 5 days, plus a single dose of oral dexamethasone 10 mg during the index ED visit, then a placebo (no active ingredient) pill daily x 4 days. Subjects in all three arms will have the option to take oral acetaminophen 975 mg every 8 hours as needed for uncontrolled pain.

Subjects will be followed up by phone at 1 day, 3 days, 7 days, and 14 days and assessed for pain, adverse events, and other outcomes. Chart review will be performed at 14 and 28 days to assess for other adverse events. All research data will be documented on standardized data collection forms.

DATA ANALYSIS

Descriptive statistics will be reported as means/medians with standard deviation/interquartile range for continuous variables and proportions with percentages for categorical variables. Differences in continuous outcome variables between the three study groups will be compared via one way ANOVA. Subsequent pairwise comparisons will utilize the Student T-test for parametric data and the Mann-Whitney U test for non-parametric data with associated 95% confidence intervals. Differences in dichotomous variables between groups will be compared via chi-squared or Fisher's exact tests, as appropriate. Primary analysis will be conducted on an intention-to-treat basis; however, per protocol sensitivity analysis is also planned. Interrater reliability for follow-up data collection from the medical record will be assessed via Cohen's kappa. p < 0.05 will be considered statistically significant.

POWER CALCULATIONS AND PLANNED SAMPLE SIZE

Power calculations are based on prior published literature on patients presenting with pain related to hip OA. Assuming an approximate baseline pain VAS mean=5/SD=2.2 and an expected mean change in numerical pain score at 72-hours change of 0.5 in the control group and 1.5 in the steroid groups, we need to enroll 59 subjects per arm to achieve 80% power at alpha=0.05. These assumptions also align with the clinically significant margin of difference in pain score (1.0) established in prior studies. Allowing for 5% attrition and need for a total enrollment equally divisible into 3 arms, we plan to enroll a total of 192 subjects (64 per arm, randomized 1:1:1).

RISKS TO SUBJECTS

While NSAIDs and glucocorticoids are very frequently administered medications, there are risks associated with their use. NSAIDs have been associated with gastric/peptic irritation/ulcers, renal adverse effects (kidney injury, electrolyte/fluid disorders, renal papillary necrosis, and interstitial nephritis) and cardiovascular adverse effects (myocardial infarction, thromboembolic events, and atrial fibrillation), as well as hepatic or hematologic effects; however, significant adverse effects from ibuprofen are rare, particularly when taken in a short course in the absence of contraindications. Ibuprofen is available over the counter without a prescription and is generally very well tolerated.

Glucocorticoids have been associated with adverse effects affecting the musculoskeletal system (osteoporosis, myopathy, osteonecrosis), endocrine system (elevated blood glucose, cushingoid features, weight gain, hirsutism/alopecia), cardiovascular system (hypertension, fluid retention, arrhythmias), and gastrointestinal system (ulcers, GIB). They are also associated with increased rates of infection and neuropsychiatric effects, such as anxiety, depression, psychosis, and sleep disturbances. However, the incidence and severity of these effects are linked to the glucocorticoid dose and duration; short courses are very commonly used in clinical practice and generally well tolerated.

There is a slight risk of the participants' privacy or confidentiality being breached. Standard precautions will be taken to ensure privacy and confidentiality are maintained during the study. There are no additional required study visits.

COSTS AND COMPENSATION

No compensation will be given to participants. There will be no research-related costs to the patient. Study medications will be provided to participants at no cost.

POTENTIAL BENEFITS TO SUBJECTS

Subjects may receive clinical benefit from the additional anti-inflammatory effect provided by glucocorticoids; however, determining the effectiveness of glucocorticoids in this clinical application is the purpose of the study. Subjects may not directly benefit from participation but may help to improve the care of patients suffering from acute OA-related pain in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute monoarticular arthritic joint pain affecting native knee, hip, or shoulder presumed to be related to osteoarthritis
* Acute pain above baseline starting less than 72 hour prior to ED visit
* Planned discharge from the ED
* History of osteoarthritis of the affected joint based on radiography performed at index visit or prior available imaging

Exclusion Criteria:

* Trauma to the affected joint within 30 days
* Injection of affected joint within 60 days
* Prior arthroplasty of the affected joint
* History of coronary artery disease, severe gastrointestinal bleeding, gastric/peptic ulcer disease, chronic kidney disease with GFR less than 30, or platelet disorders (including von Willebrand disease, hemophilia, severe thrombocytopenia with platelets less than 50 k/mcL)
* Joint pain suspected to be related to rheumatoid arthritis, gout, septic arthritis, or other non-osteoarthritis autoimmune/inflammatory/infectious arthritis
* Chronic/baseline use of glucocorticoids (greater than 5 mg daily prednisone or equivalent within previous 7 days) or NSAIDs (daily use for more than 2 days prior to presentation)
* Daily prescription opioid use or active opioid use disorder
* Illicit drug use
* Known allergy/intolerance to ibuprofen/NSAIDs, prednisone, dexamethasone, or other medication precluding ability to participate in one or more study arms
* Other contraindications to ibuprofen/NSAIDs or glucocorticoids
* Planned hospitalization from the ED
* Pregnancy
* Incarceration
* Inability to provide informed consent
* Other conditions that would preclude compliance with the study protocol and medication dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Resting Pain Score at 3 Days (Effectiveness Outcome) | 3 days (72 hours)
  Change in resting pain score from baseline at time of randomization based on subject-reported numerical resting pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 3.
Adverse Events (Safety Outcome) | 28 days
  Occurrence of adverse events reported during follow up phone calls on Day 1, 3, 7 and 14 or during chart review on Day 14 and 28, including:
  * Hyperglycemia requiring discontinuation of the study medication
  * Diabetic ketoacidosis or hospitalization for diabetes-related process
  * Bleeding events, including gastrointestinal bleeding (GIB)
  * Abdominal pain requiring discontinuation of the study medication
  * Worsening renal function requiring discontinuation of the study medication
  * Other adverse events necessitating discontinuation of study medication
  * Repeat visit to an emergency department
  * Hospitalization
  * Death

SECONDARY OUTCOMES:
Change in Resting Pain Score at 1 Day | 1 day (24 hours)
  Change in resting pain score from baseline at time of randomization based on subject-reported numerical resting pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 1.
Change in Resting Pain Score at 7 Days | 7 days
  Change in resting pain score from baseline at time of randomization based on subject-reported numerical resting pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 7.
Change in Resting Pain Score at 14 Days | 14 days
  Change in resting pain score from baseline at time of randomization based on subject-reported numerical resting pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 14.
Change in Ambulatory/Active Movement Pain Score at 1 Day | 1 day (24 hours)
  Change in ambulatory/active pain score from baseline at time of randomization based on subject-reported numerical ambulatory/active pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 1.
Change in Ambulatory/Active Movement Pain Score at 3 Days | 3 days (72 hours)
  Change in ambulatory/active pain score from baseline at time of randomization based on subject-reported numerical ambulatory/active pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 3.
Change in Ambulatory/Active Movement Pain Score at 7 Days | 7 days
  Change in ambulatory/active pain score from baseline at time of randomization based on subject-reported numerical ambulatory/active pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 7.
Change in Ambulatory/Active Movement Pain Score at 14 Days | 14 days
  Change in ambulatory/active pain score from baseline at time of randomization based on subject-reported numerical ambulatory/active pain score (0-10) for pain in the affected joint obtained during the follow up phone call on Day 14.
Use of Rescue Medication for Pain (Acetaminophen) | 14 days
  The total number of acetaminophen doses taken as needed for uncontrolled pain since discharge from the emergency department, as reported by the subject during the follow up phone call on Day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Becker, MD, Principal Investigator — WellSpan Health
Locations (1):
- WellSpan York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The study, including data collection and analysis is being conducted at a single site.

REFERENCES:
- [Background] Estee MM, Cicuttini FM, Page MJ, Butala AD, Wluka AE, Hussain SM, Wang Y. Efficacy of corticosteroids for hand osteoarthritis - a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2022 Jul 13;23(1):665. doi: 10.1186/s12891-022-05619-9. PMID 35831847
- [Background] Chou R, Pinto RZ, Fu R, Lowe RA, Henschke N, McAuley JH, Dana T. Systemic corticosteroids for radicular and non-radicular low back pain. Cochrane Database Syst Rev. 2022 Oct 21;10(10):CD012450. doi: 10.1002/14651858.CD012450.pub2. PMID 36269125
- [Background] Phillips M, Bhandari M, Grant J, Bedi A, Trojian T, Johnson A, Schemitsch E. A Systematic Review of Current Clinical Practice Guidelines on Intra-articular Hyaluronic Acid, Corticosteroid, and Platelet-Rich Plasma Injection for Knee Osteoarthritis: An International Perspective. Orthop J Sports Med. 2021 Aug 31;9(8):23259671211030272. doi: 10.1177/23259671211030272. eCollection 2021 Aug. PMID 34485586
- [Background] Juni P, Hari R, Rutjes AW, Fischer R, Silletta MG, Reichenbach S, da Costa BR. Intra-articular corticosteroid for knee osteoarthritis. Cochrane Database Syst Rev. 2015 Oct 22;2015(10):CD005328. doi: 10.1002/14651858.CD005328.pub3. PMID 26490760
- [Background] Dorleijn DMJ, Luijsterburg PAJ, Reijman M, Kloppenburg M, Verhaar JAN, Bindels PJE, Bos PK, Bierma-Zeinstra SMA. Intramuscular glucocorticoid injection versus placebo injection in hip osteoarthritis: a 12-week blinded randomised controlled trial. Ann Rheum Dis. 2018 Jun;77(6):875-882. doi: 10.1136/annrheumdis-2017-212628. Epub 2018 Mar 7. PMID 29514801
- [Background] Dossing A, Nielsen SM, Kroon FP, Balsby IM, Tarp S, Kloppenburg M, Stamp L, Haugen IK, Altman RD, Henriksen M, Boesen M, Bliddal H, Berg S, Christensen R. Comparative effectiveness of pharmacological interventions for hand osteoarthritis: a systematic review and network meta-analysis of randomised trials. RMD Open. 2023 Aug;9(3):e003030. doi: 10.1136/rmdopen-2023-003030. PMID 37734873
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149
- [Background] Long H, Liu Q, Yin H, Wang K, Diao N, Zhang Y, Lin J, Guo A. Prevalence Trends of Site-Specific Osteoarthritis From 1990 to 2019: Findings From the Global Burden of Disease Study 2019. Arthritis Rheumatol. 2022 Jul;74(7):1172-1183. doi: 10.1002/art.42089. Epub 2022 Jun 2. PMID 35233975
- [Background] Irizarry E, Restivo A, Salama M, Davitt M, Feliciano C, Cortijo-Brown A, Friedman BW. A randomized controlled trial of ibuprofen versus ketorolac versus diclofenac for acute, nonradicular low back pain. Acad Emerg Med. 2021 Nov;28(11):1228-1235. doi: 10.1111/acem.14321. Epub 2021 Jun 30. PMID 34133820
- [Background] Young SE, Bothwell JD, Walsh RM. Safely Managing Acute Osteoarthritis in the Emergency Department: An Evidence-Based Review. J Emerg Med. 2016 Dec;51(6):648-657. doi: 10.1016/j.jemermed.2016.05.052. Epub 2016 Jul 29. PMID 27480348
- [Background] Sacks JJ, Luo YH, Helmick CG. Prevalence of specific types of arthritis and other rheumatic conditions in the ambulatory health care system in the United States, 2001-2005. Arthritis Care Res (Hoboken). 2010 Apr;62(4):460-4. doi: 10.1002/acr.20041. PMID 20391499